CLINICAL TRIAL: NCT01323478
Title: A Long-term, Open-label, Flexible-dose, Extension Study Evaluating the Safety and Tolerability of [Vortioxetine] Lu AA21004 (15 and 20 mg/Day) in Patients With Major Depressive Disorder
Brief Title: Open-label Safety Extension Study of 15 and 20 mg of Vortioxetine (Lu AA21004) in Long-term Treatment of Major Depressive Disorder in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13267B; 2010-024198-38 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
Keywords: Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders; Behavioural Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Mood Disorders; Mental Disorders; Behavioral Symptoms | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)

INTERVENTIONS:
Drug: Vortioxetine (Lu AA21004) — 15 or 20 mg/day; tablets; orally
  Other Names: Brintellix

SUMMARY:
To evaluate the long-term safety and tolerability of flexible doses, 15 and 20 mg/day, of Vortioxetine over a period of 52 weeks in patients with Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

Patients who completed 8-week short-term treatment study, 13267A (NCT01140906), for Major Depressive Episode immediately prior to enrolment in this extension study

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV TR)
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication
* The patient, in the investigator's clinical judgment, has a significant risk of suicide.

Other protocol-defined inclusion and exclusion criteria applied.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Mattingly GW, Necking O, Schmidt SN, Reines E, Ren H. Long-term safety and efficacy, including anhedonia, of vortioxetine for major depressive disorder: findings from two open-label studies. Curr Med Res Opin. 2023 Apr;39(4):613-619. doi: 10.1080/03007995.2023.2178082. Epub 2023 Mar 8. PMID 36884024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients eligible to participate in Study 13267B were patients who had completed lead-in Study 13267A (NCT01140906) immediately prior to inclusion into present study, 13267B. The doses of Vortioxetine used in this long-term safety extension study were the same as those used in lead-in Study 13267A (NCT01140906).
Pre-assignment Details: The study consisted of a 52-week open-label period and a 4-week Safety Follow-up Period.
Period: Overall Study
Arm/Group | Vortioxetine 15 or 20 mg/Day
Started | 71
Completed | 47
Not Completed | 24
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 4
Not completed — Non-compliance With Study Product | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal of Consent | 1
Not completed — Administrative or Other Reasons | 8

BASELINE CHARACTERISTICS:
Population: Age and Gender: all-patients-treated set (APTS) - all patients who took at least one dose of Vortioxetine.
  Study Specific Characteristics: full-analysis set (FAS) - all 71 patients in the APTS who had at least one valid post-Baseline assessment of the MADRS total score in present study, 13267B.
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 18
MADRS: Baseline present study, 13267B [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 16.2 (10.0)
CGI-S: Baseline present study, 13267B [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 3.0 (1.3)
HAM-A: Baseline present study, 13267B [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 11.9 (6.6)
MADRS: Baseline from lead-in study 13267A (NCT01140906) [Mean (Standard Deviation); unit: units on a scale] | 31.1 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Time Frame: Baseline to end of the 4-week safety follow-up period
Population: all-patients-treated set (APTS)
Measure: Number; unit: participants
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 71
participants
  Patients With AEs | 56
  Patients With Serious AEs (SAEs) | 1
  Patients With AEs Leading to Withdrawal | 7

2. Primary Outcome: Percentage of Patients Who Withdrew Due to Intolerance to Treatment
Time Frame: Baseline to Week 52
Population: APTS
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 71
percentage of patients | 9.9

3. Secondary Outcome: Change From Baseline in MADRS Total Score After 52 Weeks of Treatment
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: full-analysis set (FAS), observed cases (OC)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 47
units on a scale | -10.9 (9.99)

4. Secondary Outcome: Change From Baseline in CGI-S Score After 52 Weeks of Treatment
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Baseline and Week 52
Population: FAS, OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 47
units on a scale | -1.49 (1.46)

5. Secondary Outcome: Change From Baseline in HAM-A Total Score After 52 Weeks of Treatment
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
Time Frame: Baseline and Week 52
Population: FAS, OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 47
units on a scale | -7.85 (7.49)

6. Secondary Outcome: Proportion of Responders at Week 52 (Response Defined as a >=50% Decrease in MADRS Total Score)
Time Frame: Baseline from lead-in study 13267A (NCT01140906) and Week 52
Population: FAS, OC
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 47
percentage of patients | 93.6

7. Secondary Outcome: Proportion of Remitters at Week 52 (Remission Defined as a MADRS Total Score <=10)
Time Frame: Baseline and Week 52
Population: FAS, OC
Measure: Number; unit: percentage of patients
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 47
percentage of patients | 80.9

8. Secondary Outcome: SDS Total Score After 52 Weeks of Treatment
Description: The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
Time Frame: Week 52
Population: FAS, OC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 34
units on a scale | 4.85 (5.84)

9. Secondary Outcome: ASEX Total Score After 52 Weeks of Treatment
Description: The Arizona Sexual Experience Scale (ASEX) is a 5-item, patient selfrated scale that evaluates a patient's recent sexual experience. Patients are asked to assess their own experience over the last week (for example, "How strong is your sex drive?", "Are your orgasms satisfying?") and respond on a 6-point scale for each item. The ASEX is used to identify individuals with sexual dysfunction. Possible total score ranges from 5 to 30, with the higher score indicating more patient sexual dysfunction.
Time Frame: Week 52
Population: APTS, OC
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 47
units on a scale | 18.60 (0.96)

10. Secondary Outcome: Risk of Suicidality Using C-SSRS Scores
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) was developed by researchers at Columbia University as a tool to systematically assess suicidal ideation and behaviour in patients during participation in a clinical study. The C-SSRS is composed of questions that address suicidal behaviour and questions that address suicidal ideation, with subquestions that assess severity. The tool was administered via an interview with the patient. Different versions of the C-SSRS are available. In this study, the Since Last Visit Version was used at all visits. In order to assess the potential relationship between Vortioxetine and suicidality more accurately and systematically, C-SSRS data were collected during the Entire Study Period.
Time Frame: Up to 52 weeks
Population: Suicidal Ideation and Behaviour Based on C-SSRS Scores by Columbia Classification Algorithm for Suicide Assessment (C-CASA) - APTS
Measure: Number; unit: participants
Arm/Group | Vortioxetine 15 or 20 mg/Day
Number analyzed (Participants) | 71
participants
  No suicidal ideation or behaviour | 67
  Any non-suicidal self-injurious behavior | 0
  Suicidal Ideation | 4
  Preparatory action towards imminent suicidal behav | 0
  Not fatal suicide attempt | 0
  Completed suicide | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 52-week open label period and 4-week safety follow-up period Other Adverse Events: 52-week open label period
Arm/Group | Vortioxetine 15 or 20 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/71
Other Adverse Events (participants affected / at risk) | 47/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 15 or 20 mg/Day (N=71)
Cholelithiasis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 15 or 20 mg/Day (N=71)
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 4
Nasopharyngitis (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 5
Accidental overdose (Injury, poisoning and procedural complications) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The primary publication must be published before any secondary publications. H. Lundbeck A/S will ensure that the authorship of all publications based on this study is in accordance with the criteria defined by the International Committee of Medical Journal Editors (ICMJE).